CLINICAL TRIAL: NCT06801808
Title: Evaluation of HMB Supplementation on Motor Performance in Sarcopenic Patients
Brief Title: HMB Supplementation and Motor Performance in Sarcopenic Patiens
Acronym: HMB-SARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000032/25
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Older adults; Nutrition; HMB
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Interventional randomized controlled pilot study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-MyO group (Experimental): Patients in G-MyO group, in addition to the pharmacological therapy routine, will take 2 sachets of Myosave per day for 8 weeks (T0-T2), followed by no product supplementation for the next 8 weeks (T2-T4)
  Interventions: Dietary Supplement: Myosave
- G-OMy group (Experimental): Patients in G-OMy group, without any changes to their pharmacological routine, will not take the product for the first 8 weeks (T0-T2) and will take 2 sachets of Myosave per day for the next 8 weeks (T2-T4)
  Interventions: Dietary Supplement: Myosave

INTERVENTIONS:
Dietary Supplement: Myosave — Nutritional supplementation with Myosave

SUMMARY:
Aging is often accompanied by the reduction and weakening of muscle mass, a condition defined as sarcopenia. According to the most recent criteria from the European Working Group on Sarcopenia in Older People, sarcopenia is considered probable when low muscle strength is documented in the patient. The diagnosis of sarcopenia is then confirmed by the presence of reduced muscle mass quantity or quality; it is classified as severe when low muscle strength, reduced muscle quantity and quality, and poor physical performance are all present. According to a recent systematic review of 130 studies, sarcopenia is estimated to affect 10-16% of older adults worldwide. Low muscle strength and rapid atrophy may also result from prolonged immobility, which is an undesirable consequence of hospitalization after illness or injury.

Approximately 65% of elderly patients experience reduced ambulatory function due to hospitalization, and between 30% and 55% report a decline in daily living activities. It has been reported that healthy older adults lose 1 kg (approximately 6%) of lean tissue in the lower limbs after 10 days of bed rest, with a corresponding 16% decline in isokinetic strength of the knee extensors. Muscle atrophy during bed rest is primarily attributed to a marked decrease in skeletal muscle protein synthesis rates, although an accelerated rate of muscle protein degradation compared to synthesis cannot be ruled out. The onset of sarcopenia is further promoted by inflammation, immunosenescence, anabolic resistance, and increased oxidative stress.

Since proper diet, physical activity, and supplementation are currently considered the fundamental pillars for the treatment and prevention of sarcopenia, the identification of a specific food for special medical purposes (AFMS) capable of slowing the progression of sarcopenia is extremely important. Treating sarcopenia also means preventing the associated negative outcomes, including lower overall and progression-free survival rates, postoperative complications, extended hospital stays in patients with various medical conditions, as well as falls and fractures, metabolic disorders, cognitive decline, and mortality in the general population.

DETAILED DESCRIPTION:
Myosave® is an AMFS formulated with a specific blend of β-hydroxy-β-methylbutyrate (HMB), sucrosomial® magnesium, sucrosomial® iron, sucrosomial® vitamin D3, sucrosomial® chromium, and amino acids, for the dietary management of sarcopenia and other conditions characterized by muscle mass loss. HMB is a metabolite of leucine that has an anabolic effect on muscles when taken in combination with physical exercise . In healthy older adults engaging in physical activity, HMB (3 g/day) consumed for 8 weeks tended to increase lean mass gain and significantly improved the percentage of body fat loss compared to the placebo group. Furthermore, daily supplementation with HMB (plus arginine and lysine) in older women over 12 weeks significantly improved function and strength. It therefore seems plausible that HMB supplementation could mitigate muscle loss in bedridden elderly patients.

Based on the existing literature, the aim of the study is to evaluate the contribution of Myosave® supplementation to motor performance, cognitive performance, fatigue, and body composition in post-bedrest sarcopenic patients.

Thirty patients of both sexes will be recruiteed, evaluated and treated at the UOC Cardiovascular Internal Medicine and the UOS Post-Acute Rehabilitation units, Fondazione Policlinico Universitario A. Gemelli IRCCS of Rome.

Patients will be divided into two groups by randomization, as specified later. One group (G-MyO), in association with the drug therapy already underway, will take 2 sachets of Myosave® per day for 8 weeks, followed by an 8-week observation period. The other group (G-OMy) will undergo an 8-week observation period first, followed by the intake of 2 sachets of Myosave® per day for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 99 years;
* Diagnosis of sarcopenia according to the criteria of the European Working Group on Sarcopenia in Older People (EWGSOP) (Cruz-Jentoft et al., 2018; Kirk et al., 2024), specifically:

  * Reduced muscle mass, assessed through bioelectrical impedance analysis (Skeletal Mass Index/height value of ≤ 7.0 kg/m² for men and ≤ 5.5 kg/m² for women);
  * Reduced muscle strength, assessed through the Hand Grip Strength Test (value < 27 kg for men and < 16 kg for women);
  * Reduced physical performance, assessed through gait speed (≤ 0.8 m/s in the 4-meter walking test) and the Short Physical Performance Battery (score ≤ 8).
* Cognitive abilities sufficient to follow simple instructions and understand the physiotherapist's guidance (assessed using the Mini Mental State Examination, with a corrected score between 22 and 27).
* Ability to walk independently or with minimal assistance;
* A history of bed rest lasting at least 5 days;
* Ability to understand and sign the informed consent form.

Exclusion Criteria:

* Presence of a known or suspected allergy/intolerance to one or more ingredients of Myosave;
* Presence of kidney or liver diseases;
* Use of anticoagulant or antiplatelet drugs;
* Presence of uncontrolled hypertension or diabetes;
* Oncological diseases, orthopedic or postural issues, presence of plantar ulcers;
* Partial or total amputation of foot segments;
* Inability to provide informed consent.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Hand grip strenght test (HGST) | Change from Baseline HGT at 8 and 16 weeks
  HGT is a test performed with a dynamometer, which goes to assess muscle strength (in kilograms). Starting with the elbow flexed to 90° the patient must squeeze the dynamometer as hard as they can at one time. Three repeated measurements are taken on each side 20 seconds apart.
  The average of the three assessments is used as the final value.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 8 and 16 weeks
  SPPB is a set of clinical tests used to assess physical performance, particularly lower extremity strenght and functional capacity in older adults. It includes three main components: balance (feet side-by-side, semitandem, and tandem positions), gait speed (time spent to walk 4m), and chair stand tests (five times chair sit-to-stand test). Each test is scored on a scale from 0 to 4, with higher scores indicating better performance. The total score ranges from 0 to 12, with higher scores reflecting better overall physical function.
Time Up&Go Test (TUG) | Change from Baseline TUG at 8 and 16 weeks
  TUG measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severely abnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from initial getting up to re-seating. Patients are compared with the mean time of adults in their age group, 60 to 69, 70 to 79, and 80 to 99 years of age.
Timed 25 Foot Walk (T25FW) | Change from Baseline T25FW at 8 and 16 weeks
  The T25FW is a performance- based test used to measuere walking speed and mobility. The individuals is asked to walk a distance of 25 feet (approximately 7.62 meters) as quickly and safely as possible, with or without the use of assistive devices. The time taken to complete the walk is recorded, and the test is typically performed twice to ensure accuracy.
Trial Making Test (TMT) | Change from Baseline TMT at 8 and 16 weeks
  The TMT measueres flexibility of thinking on a visual-motor sequencing task. It consist of two parts, A and B where 25 circles distributed over a sheet paper. In part A, the circles are numbered 1-25, and the patient should draw lines to connect the numbers in ascending order. In part B, the circles include both numbers (1-13) and letters (A-L9: as pattern, but with the added task of alternating between the numebrs and lettes (i.e., 1-A-2-b-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, deficient> 78 seconds, Rule of Thumb most in 90 seconds. Trial B: Averange 75 seconds, deficient> 273 seconds, Rule of Thumb most in 3 minutes
Symbol Digit Modalities Test (SDMT) | Change from Baseline SDMT at 8 and 16 weeks
  The SDMT is a neuropsycological test used to assess cogntive processing speed, attention, and visual-motor coordination. The test involves matching symbols to corresponding numbers based on a key, and participants must quickly and accurately pair the symbols with the correct numbers within a set time limit.
  The test evaluates attention, working memory, and mental flexibility. A higher score indicates better cognitive processing speed and accuracy.
Stroop colour Word Test (SCWT) | Change from Baseline SCWT 8 and 16 weeks
  The SCWT is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task, to name colors in the second and third tasks. It is necessary to mark both any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Hospital Anxiety and depression scale (HADS) | Change from Baseline SCWT 8 and 16 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a tool used to check for symptoms of anxiety and depression, especially in hospital patients. It has 14 questions, 7 for anxiety and 7 for depression. Each question is scored from 1 to 4.
Modified Fatigue Impact scale (MFIS) | Change from Baseline SCWT 8 and 16 weeks
  The Modified Fatigue Impact Scale (MFIS) is a tool used to assess the impact of fatigue on a person's physical, cognitive, and psychosocial functioning. It consists of 21 items, each scored from 0 (never) to 4 (almost always), with higher scores indicating greater fatigue impact. The scale is divided into three subscales: physical, cognitive, and psychosocial, providing a comprehensive measure of how fatigue affects daily life.
EuroQoL-5D (EQ-5D) | Change from Baseline SCWT 8 and 16 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Mini Nutritional Assessment- short Form (MNA-SF) | Change from Baseline SCWT 8 and 16 weeks
  The Mini Nutritional Assessment - Short Form (MNA-SF) is a screening tool used to quickly evaluate the risk of malnutrition in older adults. It consists of 6 questions covering aspects such as weight loss, appetite, mobility, psychological stress, and body mass index (BMI) or calf circumference. Scores range from 0 to 14, with 12-14 indicating normal nutrition, 8-11 at risk of malnutrition, and 0-7 indicating malnutrition.
SARC-F | Change from Baseline SCWT 8 and 16 weeks
  The SARC-F is a simple screening tool used to identify individuals at risk of sarcopenia. It consists of 5 questions assessing strength, assistance with walking, rising from a chair, climbing stairs, and falls. Each item is scored from 0 to 2, with a total score ranging from 0 to 10. A score of 4 or higher suggests a risk of sarcopenia and the need for further assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia MD Giovannini, phD, Principal Investigator — Fondazione Policlinico Iniversitario A.Gemelli, IRCSS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy